CLINICAL TRIAL: NCT01862263
Title: A Multicenter, Double-Blind, Randomized, Parallel-Group Placebo-Controlled Study to Compare the Effect of 13-Week Treatment With Vildagliptin as Add-On Therapy to Improve Glucose Variability in Type 2 Diabetes Mellitus Patients Inadequately Controlled With Insulin.
Brief Title: Effect of 13-Week Treatment With Vildagliptin as Add-On Therapy to Improve Glucose Variability in Type II Diabetes
Acronym: VIDA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLAF237AMX01
Record Dates: First submitted 2013-05-22; First posted 2013-05-24 (Estimated); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes,; Type 2 diabetes,; Diabetes mellitus,; insulin,
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance | interventions — Vildagliptin; Insulin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vildagliptin (Experimental): Vildagliptin 50 mg twice daily (bid) + Insulin 20 to 40 IU/day
  Interventions: Drug: Vildagliptin; Drug: Insulin
- Placebo (Placebo Comparator): Insulin 20 to 40 IU/day + Vildagliptin Placebo twice daily (bid)
  Interventions: Drug: Insulin; Drug: Placebo

INTERVENTIONS:
Drug: Vildagliptin — Orally active and highly selective inhibitor of DPP-4
  Arms: Vildagliptin
Drug: Insulin — Long- acting human insulin analog indicated to improve glycemic control
Drug: Placebo — Matching placebo of vildagliptin
  Arms: Placebo

SUMMARY:
The purpose of the study is to assess if the addition of vildagliptin as add-on therapy improves glucose variability in type 2 diabetes mellitus (T2DM) patients inadequately controlled with insulin, with special emphasis in hypoglycemic episodes measured by continuous glucose monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent read and signed before any protocol procedure.
2. Free will to sign the informed consent.
3. Male and female between 18 and 80 years. If female, patient must be non-fertile or of childbearing potential using a medically approved birth control method.
4. Type 2 diabetes mellitus
5. Patient under insulin treatment within 3 years with stable insulin NPH (Neutral ProtamineHagedorn) regimen at dose of at least 20 UI/day up to 40 UI/day for a minimum of 4 weeks prior to enrolment, only NPH and glargine insulin are allowed.
6. HbA1c between 7.5 to 9%.
7. Fasting plasma glucose (FPG) less than 270 mg/dL.
8. Body mass index (BMI) between 20 to 35 kg/m2.
9. Free willing to take the vildagliptin tablets during the study.

Exclusion Criteria

1. Pregnant or lactating female or without birth control method if of childbearing potential.
2. Type 1 diabetes, diabetes that is a result of pancreatic injury, or secondary forms of diabetes, e.g., Cushing's syndrome.
3. Acute cardiovascular complications or metabolic complications within the past 4 months.
4. History cerebrovascular disease during the last year.
5. History of Torsades de Points, ventricular tachycardia or ventricular fibrillation.
6. Ischemic heart disease (e.g. myocardial infarction, unstable angina, coronary artery bypass surgery).
7. Congestive heart failure requiring pharmacologic treatment.
8. Any known serious heart condition.
9. ALT and/or AST greater than three times the upper limit of the normal range.
10. Serum creatinine levels greater than 1.5 mg/dL
11. Malignancy including leukemia and lymphoma within the last 5 years

Other inlcusion/exclusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2013-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with hyperglycemic events evaluated with CGM | At 13 weeks
  An hypoglycemic event is defined as any continuous glucose monitoring (CGM) measurement less than 60 mg/dL and a hyperglycemic is define as any CGM greater than 140 mg/dL.

SECONDARY OUTCOMES:
Number of hypoglycemia and/or hyperglycemia measured by CGM | 13 weeks
  An episode of hypoglycemia is defined as any value of glucose under 60 mg/dL, an episode of hyperglycemia is defined as any value of glucose above 140mg/dL measured by CGM.
Area under the curve (AUC 0-24) of the excursions of glucose values below 60 mg/dl per day | 0 to 24 hours daily for week 1, 4 and 13
  Duration and intensity of hypoglycemic episodes, measured as area under the curve (AUC 0-24) of the excursions of glucose values below 60 mg/dl per day, measured by continuous glucose monitoring
Average of insulin units per day administered during the study | 13 weeks
  Change from baseline
Changes from the baseline in Lipid Profile | Baseline, 13 weeks
  Lipid Profile will include total cholesterol, HDL cholesterol, LDL cholesterol, VLDL cholesterol
Change from baseline in Body weight | Baseline, 13 weeks
  Weight will be measured on Kg.
Change from baseline in Blood pressure (BP), | Baseline, 13 weeks
  BP will be mesured on mmHg
Change from baseline in Fasting plasma glucose (FPG), | Baseline, 13 weeks
  FPG will be measured on mg/dL
Change from baseline in Hemoglobin A1C (HbA1c) | Baseline, 13 weeks
  HbA1c will be measured on %
Change from baseline in Creatinine | Baseline, 13 weeks
  Creatinine will be measured on mg/dL
Change from baseline in C-peptide | Baseline, 13 weeks
  C-Peptide will be measured on microIU/mL
Changes from baseline in alanine aminotransferase (ALT)/aspartate aminotransferase (AST) | Baseline, 13 week
  ALT/AST will be measured on ratio.
Changes from baseline in Direct bilirubin | Baseline, 13 weeks
  Bilirubin will be measure on mg/dL
Changes from baseline in Body Mass Index (BMI) | Baseline, 13 weeks
Number of patients with adverse events, serious adverse events and death as evaluation of safety and tolerability of coadministration of vildagliptin with insulin | 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- Mexico (8):
  - Novartis Investigative Site, Celaya, Guanajuato
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, Monterrey, Nuevo León
  - Novartis Investigative Site, Cancún, Quintana Roo
  - Novartis Investigative Site, Culiacán, Sinaloa
  - Novartis Investigative Site, Metepec, State of Mexico
  - Novartis Investigative Site, Puebla City